CLINICAL TRIAL: NCT02873598
Title: A Dose Escalation Trial of Stereotactic Body Radiotherapy (SBRT) After Induction Chemotherapy for Locally Advanced Pancreatic Cancer
Brief Title: A Dose Escalation Trial of SBRT After Induction Chemotherapy for Locally Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 16-1139.cc
Record Dates: First submitted 2016-08-08; First posted 2016-08-19 (Estimated); Results first posted 2022-10-13 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Pancreatic Cancer
Keywords: Induction Chemotherapy; Stereotactic Body Radiotherapy (SBRT); Dose Escalation; Locally Advanced Pancreatic Cancer (LAPC); Maximum Tolerated Dose (MTD)
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — folfirinox; Gemcitabine; Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Intervention Model Description: Dose escalation will start with dose level 1 (9 Gy x 3 fractions) and increase by 1 Gy per fraction at each dose level, dose level 2 will be 10 Gy x 3 fractions and dose level 3 will be 11 Gy x 3 fractions.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- FOLFIRINOX or gemcitabine/abraxane followed by SBRT Dose level 1 (Experimental): SBRT will be administered in 3 fractions, every other day, on an outpatient basis, following chemotherapy with either FOLFIRINOX or gemcitabine/abraxane. Dose level 1- 9 Gy x 3 fractions.
  Interventions: Drug: FOLFIRINOX or gemcitabine/abraxane; Radiation: SBRT
- FOLFIRINOX or gemcitabine/abraxane followed by SBRT Dose level 2 (Experimental): SBRT will be administered in 3 fractions, every other day, on an outpatient basis, following chemotherapy with either FOLFIRINOX or gemcitabine/abraxane. Dose level 2 -10 Gy x 3 fractions
  Interventions: Drug: FOLFIRINOX or gemcitabine/abraxane; Radiation: SBRT
- FOLFIRINOX or gemcitabine/abraxane followed by SBRT Dose level 3 (Experimental): SBRT will be administered in 3 fractions, every other day, on an outpatient basis, following chemotherapy with either FOLFIRINOX or gemcitabine/abraxane. Dose level 3 - 11 Gy x 3 fractions.
  Interventions: Drug: FOLFIRINOX or gemcitabine/abraxane; Radiation: SBRT

INTERVENTIONS:
Drug: FOLFIRINOX or gemcitabine/abraxane — Patients will have received induction chemotherapy for 3+ months with either FOLFIRINOX or gemcitabine/abraxane with at least stable disease.
  Other Names: nab-paclitaxel
Radiation: SBRT — After completion of induction chemotherapy, stereotactic body radiation therapy (SBRT) will be administered in 3 fractions, every other day, on an outpatient basis. Dose escalation will start with dose level 1 (9 Gy x 3 fractions) and increase by 1 Gy per fraction at each dose level, dose level 2 will be 10 Gy x 3 fractions and dose level 3 will be 11 Gy x 3 fractions.

SUMMARY:
This is a dose escalation trial to evaluate the safety of stereotactic body radiotherapy (SBRT) delivered in 3 fractions for patients with locally advanced pancreatic cancer (LAPC) who have received induction chemotherapy (FOLFIRINOX or gemcitabine and nab-paclitaxel).

DETAILED DESCRIPTION:
This is a phase I study, with an expansion cohort, of up to 34 patients to identify the maximum tolerated dose (MTD) of a 3-fraction regimen of stereotactic body radiotherapy (SBRT) for locally-advanced pancreatic cancer patients who have not developed distant progression following induction chemotherapy (FOLFIRINOX or gemcitabine and nab-paclitaxel) as per standard of care. After completion of induction chemotherapy, stereotactic body radiotherapy SBRT will be administered in 3 fractions, every other day, on an outpatient basis. Dose escalation will start with dose level 1 (9 Gy x 3 fractions) and increase by 1 Gy per fraction at each dose level, dose level 2 will be 10 Gy x 3 fractions and dose level 3 will be 11 Gy x 3 fractions.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytopathologically confirmed adenocarcinoma of the pancreas.
2. Locally advanced, unresectable pancreatic cancer as confirmed by the multidisciplinary input from a hepatobiliary surgeon and as defined on CT as having tumor abutment of >180° (> 50%) of the circumference of the superior mesenteric artery (SMA) or celiac axis, unreconstructable superior mesenteric vein (SMV) or portal vein (PV) involvement.
3. No evidence of distant metastasis either prior to or after induction chemotherapy.
4. Completion of at least 3 months, but no more than 6 months of standard induction chemotherapy for LAPC, which may include FOLFIRINOX or gemcitabine and nab-paclitaxel, preferably within 2-4 weeks but no longer than 8 weeks.
5. Pancreatic tumor size ≤ 5 cm.
6. Age ≥18 years.
7. ECOG 0-1.
8. Patients must have acceptable organ and marrow function as defined below:

   * Leukocytes >3,000/µL
   * Absolute neutrophil count >1,500/µL
   * Platelets >70,000/µL
   * Total bilirubin Within 2 x upper limit of normal
   * AST (SGOT)/ALT (SGPT) <2.5 x institutional upper limit of normal
   * Creatinine Within 1.5 x upper limit of normal OR
   * Creatinine clearance >60 mL/min for patients with creatinine levels above institutional normal
9. Ability to understand and follow the breathing instructions involved in the respiratory gating procedure or to tolerate compression sufficient to reduce fiducial motion to <= 5mm.
10. Ability to understand and the willingness to sign a written informed consent document.
11. Residual or on-going ≥ Grade 3 treatment-related toxicity from previous chemotherapy

Exclusion Criteria:

1. Patients who have had prior abdominal radiotherapy.
2. Patients receiving any investigational agents.
3. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
4. Contraindication to IV contrast
5. Patients in which iodine contrast is contraindicated.
6. Pregnant and breastfeeding women are excluded. Women of child-bearing potential who are unwilling or unable to use an acceptable method of birth control to avoid pregnancy for the entire study period and for up to 4 weeks after the study are excluded. This applies to any woman who has experienced menarche and who has not undergone successful surgical sterilization or is not postmenopausal (defined as amenorrhea for at least 12 consecutive months, or women on hormone replacement therapy with serum FSH levels greater than 35 mIU/mL. A negative urine or serum pregnancy test must be obtained within 14 days prior to the start of study therapy in all women of child-bearing potential. Male subjects must also agree to use effective contraception for the same period as above.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-11-17 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2022-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sana Karam, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- FOLFIRINOX or Gemcitabine/Abraxane Followed by SBRT Dose 1: SBRT will be administered in 3 fractions, every other day, on an outpatient basis, following chemotherapy with either FOLFIRINOX or gemcitabine/abraxane. Dose level 1 - 9 Gy x 3 fractions.
  FOLFIRINOX or gemcitabine/abraxane: Patients will have received induction chemotherapy for 3+ months with either FOLFIRINOX or gemcitabine/abraxane with at least stable disease.
  SBRT: After completion of induction chemotherapy, stereotactic body radiation therapy (SBRT) will be administered in 3 fractions, every other day, on an outpatient basis. Dose escalation will start with dose level 1 (9 Gy x 3 fractions) and increase by 1 Gy per fraction at each dose level, dose level 2 will be 10 Gy x 3 fractions and dose level 3 will be 11 Gy x 3 fractions.
- FOLFIRINOX or Gemcitabine/Abraxane Followed by SBRT Dose 2: SBRT will be administered in 3 fractions, every other day, on an outpatient basis, following chemotherapy with either FOLFIRINOX or gemcitabine/abraxane. Dose level 2 - 10 Gy x 3 fractions.
  FOLFIRINOX or gemcitabine/abraxane: Patients will have received induction chemotherapy for 3+ months with either FOLFIRINOX or gemcitabine/abraxane with at least stable disease.
  SBRT: After completion of induction chemotherapy, stereotactic body radiation therapy (SBRT) will be administered in 3 fractions, every other day, on an outpatient basis. Dose escalation will start with dose level 1 (9 Gy x 3 fractions) and increase by 1 Gy per fraction at each dose level, dose level 2 will be 10 Gy x 3 fractions and dose level 3 will be 11 Gy x 3 fractions.
- FOLFIRINOX or Gemcitabine/Abraxane Followed by SBRT Dose 3: SBRT will be administered in 3 fractions, every other day, on an outpatient basis, following chemotherapy with either FOLFIRINOX or gemcitabine/abraxane. Dose level 3 - 11 Gy x 3 fractions.
  FOLFIRINOX or gemcitabine/abraxane: Patients will have received induction chemotherapy for 3+ months with either FOLFIRINOX or gemcitabine/abraxane with at least stable disease.
  SBRT: After completion of induction chemotherapy, stereotactic body radiation therapy (SBRT) will be administered in 3 fractions, every other day, on an outpatient basis. Dose escalation will start with dose level 1 (9 Gy x 3 fractions) and increase by 1 Gy per fraction at each dose level, dose level 2 will be 10 Gy x 3 fractions and dose level 3 will be 11 Gy x 3 fractions.
Period: Overall Study
Arm/Group | FOLFIRINOX or Gemcitabine/Abraxane Followed by SBRT Dose 1 | FOLFIRINOX or Gemcitabine/Abraxane Followed by SBRT Dose 2 | FOLFIRINOX or Gemcitabine/Abraxane Followed by SBRT Dose 3
Started | 5 | 5 | 4
Completed | 5 | 5 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- FOLFIRINOX or Gemcitabine/Abraxane Followed by SBRT Dose Level 1: SBRT will be administered in 3 fractions, every other day, on an outpatient basis, following chemotherapy with either FOLFIRINOX or gemcitabine/abraxane. Dose level 1 - 9 Gy x 3 fractions.
  FOLFIRINOX or gemcitabine/abraxane: Patients will have received induction chemotherapy for 3+ months with either FOLFIRINOX or gemcitabine/abraxane with at least stable disease.
  SBRT: After completion of induction chemotherapy, stereotactic body radiation therapy (SBRT) will be administered in 3 fractions, every other day, on an outpatient basis. Dose escalation will start with dose level 1 (9 Gy x 3 fractions) and increase by 1 Gy per fraction at each dose level, dose level 2 will be 10 Gy x 3 fractions and dose level 3 will be 11 Gy x 3 fractions.
- FOLFIRINOX or Gemcitabine/Abraxane Followed by SBRT Dose Level 2: SBRT will be administered in 3 fractions, every other day, on an outpatient basis, following chemotherapy with either FOLFIRINOX or gemcitabine/abraxane. Dose level 2 - 10 Gy x 3 fractions.
  FOLFIRINOX or gemcitabine/abraxane: Patients will have received induction chemotherapy for 3+ months with either FOLFIRINOX or gemcitabine/abraxane with at least stable disease.
  SBRT: After completion of induction chemotherapy, stereotactic body radiation therapy (SBRT) will be administered in 3 fractions, every other day, on an outpatient basis. Dose escalation will start with dose level 1 (9 Gy x 3 fractions) and increase by 1 Gy per fraction at each dose level, dose level 2 will be 10 Gy x 3 fractions and dose level 3 will be 11 Gy x 3 fractions.
- Total: Total of all reporting groups
Arm/Group | FOLFIRINOX or Gemcitabine/Abraxane Followed by SBRT Dose Level 1 | FOLFIRINOX or Gemcitabine/Abraxane Followed by SBRT Dose Level 2 | FOLFIRINOX or Gemcitabine/Abraxane Followed by SBRT Dose Level 3 | Total
Number analyzed (Participants) | 5 | 5 | 4 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 2 | 5
  >=65 years | 3 | 4 | 2 | 9
Age, Continuous [Median (Full Range); unit: years] | 67 [53 to 73] | 68 [58 to 79] | 55 [52 to 79] | 67 [52 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 2 | 10
  Male | 2 | 0 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 4 | 14
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 5 | 5 | 4 | 14
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 4 | 14

OUTCOME MEASURES:

1. Primary Outcome: The Maximum Tolerated Dose (MTD) of Stereotactic Body Radiotherapy (SBRT) in Locally Advanced Pancreatic Cancer (LAPC) Patients Who Have Not Developed Distant Progression After Induction Chemotherapies.
Description: This will be accomplished by the standard 3+3 dose escalation design. Dose limiting toxicities (DLT) are defined by ≥ Grade 3 treatment-related GI toxicity within 3 months of SBRT. These include: (1) Bowel (includes bowel perforation, obstruction, or hemorrhage) and (2) Stomach (bleeding ulcer, perforation) as determined by imaging or endoscopic evaluation.
Time Frame: Up to 3 months
Measure: Number; unit: grey
Groups:
- FOLFIRINOX or Gemcitabine/Abraxane Followed by SBRT: SBRT will be administered in 3 fractions, every other day, on an outpatient basis, following chemotherapy with either FOLFIRINOX or gemcitabine/abraxane
  FOLFIRINOX or gemcitabine/abraxane: Patients will have received induction chemotherapy for 3+ months with either FOLFIRINOX or gemcitabine/abraxane with at least stable disease.
  SBRT: After completion of induction chemotherapy, stereotactic body radiation therapy (SBRT) will be administered in 3 fractions, every other day, on an outpatient basis. Dose escalation will start with dose level 1 (9 Gy x 3 fractions) and increase by 1 Gy per fraction at each dose level, dose level 2 will be 10 Gy x 3 fractions and dose level 3 will be 11 Gy x 3 fractions.
Arm/Group | FOLFIRINOX or Gemcitabine/Abraxane Followed by SBRT
Number analyzed (Participants) | 14
grey | 33

2. Secondary Outcome: Local Control
Description: Local control (LC) will be measured from completion of SBRT to the time of identification of any local progression by imaging or surgical exploration. The pattern of patients experiencing local, distant or local with distant failure will be estimated using competing risks method.
Time Frame: Up to 5 years
Reporting Status: Not Posted

3. Secondary Outcome: Progression Free Survival
Description: Progression free survival (PFS) will be measured from completion of SBRT to the time of tumor progression or death due to any cause. PFS will be estimated using the method of Kaplan and Meier.
Time Frame: Up to 5 years
Reporting Status: Not Posted

4. Secondary Outcome: Overall Survival
Description: Overall survival (OS) will be measured from completion of SBRT until death due to any cause. OS will be estimated using the method of Kaplan and Meier.
Time Frame: Up to 5 years
Reporting Status: Not Posted

5. Secondary Outcome: Small Intestine Changes
Description: Investigators will measure changes in the perfusion/permeability related parameters of peripancreatic small intestine before, during and after SBRT for patients using pCT and correlating these changes with the development of gastrointestinal toxicity such as duodenal ulcers, strictures, or enteritis. Patients will undergo baseline, post-first-fraction SBRT and post-treatment CT scans.
Time Frame: 6 weeks after SBRT
Reporting Status: Not Posted

6. Secondary Outcome: Vascular and Cellular Changes
Description: Investigators will measure changes in diffusion and perfusion/permeability by using perfusion CT derived parameters that can predict treatment response and to assess any correlation between these perfusion CT derived parameters and local control and progression-free survival
Time Frame: 6 weeks after SBRT
Reporting Status: Not Posted

7. Secondary Outcome: Quality of Life (QOL)
Description: The primary objective of the QOL study is to document the patient's experience of treatment for locally advanced pancreatic cancer by examining global QOL, physical symptoms, physical functioning and emotional well-being at baseline, during treatment, and after treatment. QOL measures including EORTC-QLQ-C30 questionnaire and the Pancreatic Cancer subscale (EORTC-PAN26) will be assessed 14 days prior to SBRT (Time 0), 10-12 weeks after SBRT (Time 1), and 6 months after SBRT (Time 2). The primary QOL endpoints include the EORTC global QOL, physical symptoms, physical functioning and emotional well-being.
Time Frame: 6 months after SBRT
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 24 months
Groups:
- FOLFIRINOX or Gemcitabine/Abraxane Followed by SBRT Dose Level 1: SBRT will be administered in 3 fractions, every other day, on an outpatient basis, following chemotherapy with either FOLFIRINOX or gemcitabine/abraxane. Dose level 1 - 9 Gy x 3 fractions
  FOLFIRINOX or gemcitabine/abraxane: Patients will have received induction chemotherapy for 3+ months with either FOLFIRINOX or gemcitabine/abraxane with at least stable disease.
  SBRT: After completion of induction chemotherapy, stereotactic body radiation therapy (SBRT) will be administered in 3 fractions, every other day, on an outpatient basis. Dose escalation will start with dose level 1 (9 Gy x 3 fractions) and increase by 1 Gy per fraction at each dose level, dose level 2 will be 10 Gy x 3 fractions and dose level 3 will be 11 Gy x 3 fractions.
- FOLFIRINOX or Gemcitabine/Abraxane Followed by SBRT Dose Level 2: SBRT will be administered in 3 fractions, every other day, on an outpatient basis, following chemotherapy with either FOLFIRINOX or gemcitabine/abraxane. Dose level 2 - 10 Gy x 3 fractions
  FOLFIRINOX or gemcitabine/abraxane: Patients will have received induction chemotherapy for 3+ months with either FOLFIRINOX or gemcitabine/abraxane with at least stable disease.
  SBRT: After completion of induction chemotherapy, stereotactic body radiation therapy (SBRT) will be administered in 3 fractions, every other day, on an outpatient basis. Dose escalation will start with dose level 1 (9 Gy x 3 fractions) and increase by 1 Gy per fraction at each dose level, dose level 2 will be 10 Gy x 3 fractions and dose level 3 will be 11 Gy x 3 fractions.
- FOLFIRINOX or Gemcitabine/Abraxane Followed by SBRT Dose Level 3: SBRT will be administered in 3 fractions, every other day, on an outpatient basis, following chemotherapy with either FOLFIRINOX or gemcitabine/abraxane. Dose level 3 - 1Gy x 3 fractions
  FOLFIRINOX or gemcitabine/abraxane: Patients will have received induction chemotherapy for 3+ months with either FOLFIRINOX or gemcitabine/abraxane with at least stable disease.
  SBRT: After completion of induction chemotherapy, stereotactic body radiation therapy (SBRT) will be administered in 3 fractions, every other day, on an outpatient basis. Dose escalation will start with dose level 1 (9 Gy x 3 fractions) and increase by 1 Gy per fraction at each dose level, dose level 2 will be 10 Gy x 3 fractions and dose level 3 will be 11 Gy x 3 fractions.
Arm/Group | FOLFIRINOX or Gemcitabine/Abraxane Followed by SBRT Dose Level 1 | FOLFIRINOX or Gemcitabine/Abraxane Followed by SBRT Dose Level 2 | FOLFIRINOX or Gemcitabine/Abraxane Followed by SBRT Dose Level 3
All-Cause Mortality (participants affected / at risk) | 4/5 | 3/5 | 4/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/5 | 1/4
Other Adverse Events (participants affected / at risk) | 4/5 | 3/5 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOLFIRINOX or Gemcitabine/Abraxane Followed by SBRT Dose Level 1 (N=5) | FOLFIRINOX or Gemcitabine/Abraxane Followed by SBRT Dose Level 2 (N=5) | FOLFIRINOX or Gemcitabine/Abraxane Followed by SBRT Dose Level 3 (N=4)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Anorexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOLFIRINOX or Gemcitabine/Abraxane Followed by SBRT Dose Level 1 (N=5) | FOLFIRINOX or Gemcitabine/Abraxane Followed by SBRT Dose Level 2 (N=5) | FOLFIRINOX or Gemcitabine/Abraxane Followed by SBRT Dose Level 3 (N=4)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anorexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2)
dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
fatigue (General disorders) | 2 (3) | 1 (3) | 1 (1)
flank pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
gastroinstestinal disorder (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 2 (2) | 1 (2) | 2 (4)
non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
vomitting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
weight loss (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-04-06): https://cdn.clinicaltrials.gov/large-docs/98/NCT02873598/Prot_SAP_ICF_000.pdf